CLINICAL TRIAL: NCT06672874
Title: Fermented Papaya and Driving Simulator Older Adult Study
Acronym: FPP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Osato Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202401429
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Fermented Papaya; Driving Simulator; Older Adults
MeSH Terms: interventions — fermented papaya preparation

STUDY DESIGN:
Intervention Model Description: All participants in this single-group study will receive the same intervention, Fermented Papaya Preparation (FPP). Each participant will serve as their own control, allowing comparisons between their baseline (pre-FPP) driving performance and subsequent assessments following FPP administration. Participants will complete three assessments in a high-fidelity driving simulator at baseline, short-term (within 24 hours post-FPP), and long-term (after 8 weeks of FPP use) to evaluate changes in cognitive functions and driving performance over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fermented Papaya Preparation (FPP) Intervention Arm (Experimental): Participants in this single-arm study will receive Fermented Papaya Preparation (FPP), administered as a 3-gram dose taken three times daily (morning, afternoon, and evening) for 8 weeks. Assessments will be conducted at three time points: baseline, within 24 hours after initial FPP administration (short-term), and after 8 weeks (long-term). This arm investigates the association between FPP and driving performance, focusing on cognitive and psychomotor functions such as attention, memory, reaction time, and executive function using a high-fidelity driving simulator.
  Interventions: Dietary Supplement: Fermented Papaya Preparation (FPP)

INTERVENTIONS:
Dietary Supplement: Fermented Papaya Preparation (FPP) — Fermented Papaya Preparation (FPP) is administered in this study as a dietary supplement aimed at assessing its potential benefits for cognitive function and driving performance in older adults. Participants consume FPP as a 3-gram powder dose taken orally three times daily (morning, afternoon, evening) for a total of 8 weeks. FPP is known for its antioxidant and anti-inflammatory properties, which may influence cognitive domains essential for safe driving, such as attention, memory, reaction time, and executive function. This intervention is specifically designed to explore FPP's potential impact on reducing driving errors and improving psychomotor skills in a high-fidelity driving simulation environment.

SUMMARY:
Yes, this additional detail will refine the original template content to emphasize the study's specific aims and hypotheses. Here's an updated version:

The goal of this clinical trial is to assess if Fermented Papaya Preparation (FPP) can enhance driving performance and reduce driving errors in community-dwelling older adults aged 70-80, who serve as their own controls. The main questions it aims to answer are:

Does FPP reduce the total number of driving errors, particularly those related to psychomotor performance? Does FPP improve driving-related cognitive functions, such as divided attention, working memory, reaction time, and executive function? How do FPP dosage, timing, and acute effects impact driving performance in adults aged 65 and older?

Participants will:

Consume three doses of FPP (3 grams per dose) within 24 hours, with the final dose administered before the simulator driving test.

Complete a high-fidelity driving simulation to assess the association between FPP use and driving errors that predict on-road performance.

Undergo baseline and post-FPP cognitive assessments to compare psychomotor performance and cognitive functions after FPP administration.

DETAILED DESCRIPTION:
This study, titled "Fermented Papaya and Driving Simulator Older Adult Study," investigates the association between Fermented Papaya Preparation (FPP) and driving performance in adults aged 70-80 using a high-fidelity driving simulator. With the aging population growing and driving safety as a critical issue among older adults, this study aims to determine whether FPP-a known antioxidant with anti-inflammatory properties-can enhance cognitive functions essential for safe driving, including attention, working memory, reaction time, and executive functions.

Participants will undergo three driving assessments in the simulator: a baseline test, a short-term follow-up (within 24 hours after FPP administration), and a long-term follow-up at 8 weeks. Each participant acts as their own control, providing comparative data on FPP's effects over time. The primary endpoints include reductions in driving errors associated with psychomotor performance and improvements in divided attention and executive functions.

Technical Aspects and Measures:

Simulator Setup and Scenario: The RTI high-fidelity simulator used in this study provides a realistic and controlled driving environment, replicating common on-road scenarios such as lane changes, reactions to environmental cues, and avoidance maneuvers. Scenarios are randomized to control for learning effects.

Visual and Cognitive Testing: Standardized tests, such as the Montreal Cognitive Assessment and the Useful Field of View, will measure baseline cognitive abilities and potential changes following FPP administration.

Simulator Sickness Management: To ensure comfort, a simulator sickness protocol is in place, including pre-study dietary recommendations and a controlled lab environment with ventilation and temperature settings.

This study could yield significant data on FPP's impact on driving skills, supporting the potential for nutraceutical interventions in promoting driving safety and independence among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 70 and 80 years.
* Community-dwelling and independent in daily living activities.
* Holds a valid driver's license and has driven in the last 3 months.
* Proficient in reading, writing, and speaking English.
* Physically able to participate in a driving simulation.
* Willing to comply with the study requirements, including FPP dosing and simulator sessions.

Exclusion Criteria:

* Currently taking psychoactive medications.
* Diagnosed with a physical disability that impairs driving ability.
* History of upper extremity amputation or right lower extremity amputation.
* Scores below 18/30 on the Montreal Cognitive Assessment (MoCA).
* Exhibits symptoms of severe simulator sickness after an initial test session.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Driving Errors Related to Cognitive Functions | Baseline, within 24 hours post-FPP administration, and at 8-week follow-up.
  The primary outcome measure for this study is the reduction in total driving errors in a high-fidelity driving simulator, with a focus on errors related to cognitive functions essential for safe driving, such as divided attention, reaction time, working memory, and executive function. This outcome will assess whether Fermented Papaya Preparation (FPP) impacts cognitive and psychomotor performance related to driving safety.

CONTACTS AND LOCATIONS:
Overall Officials: Sherrilene Classen, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- UF Smarthouse, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided